CLINICAL TRIAL: NCT00953797
Title: Role of EECP Therapy in Patients With Resistant Hypertension
Brief Title: Role of Enhanced External Counterpulsation (EECP) Therapy in Patients With Resistant Hypertension
Acronym: EECP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Darshak Karia, MD, Director of Heart Failure Services, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN4112
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
Keywords: Resistant Hypertension; Endothelial dysfunction; Enhanced External Counterpulsation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Enhanced External Counterpulsation — A non-invasive method currently used for the treatment of ischemic coronary disease. During EECP therapy three compressive pneumatic cuffs are wrapped around the calves, lower thighs, and upper thighs. The cuffs inflate sequentially during diastole causing retrograde aortic flow, and increased venous return. At end diastole, the cuffs rapidly deflate resulting in unloading of the left ventricle and a decrease in systolic blood pressure.

SUMMARY:
High Blood Pressure or Hypertension is one of the main causes of stroke, heart disease, heart attack and kidney disease. Traditionally physicians use diet and lifestyles change and medications to control patient's blood pressure. There are however, some patients whose blood pressures are difficult to control and their blood pressure remains elevated despite multiple medications. When blood pressure remains above goal (greater then 140/90 or greater then 130/80 mmHg in patients with diabetes or kidney disease) despite 3 or more blood pressure medications, the investigators call it "Resistant Hypertension".

Enhanced External Counterpulsation (EECP) is a new method of treatment currently used in people with heart disease and chest pain. EECP therapy uses three sets of balloon like cuffs that are wrapped to the calves, lower thighs, and upper thighs. These cuffs inflate and deflate with every heart beat, causing increased blood return to the heart and better blood flow. It has also been found to improve the function of endothelial cells, a type of cells that lines the wall of blood vessel through out the body which helps to regulate and maintain blood pressure. This leads us to believe that EECP therapy, although not used at present for treating patients with Resistant Hypertension, may be useful in decreasing blood pressure.

DETAILED DESCRIPTION:
Hypertension is a major cause and contributor to stroke, heart and kidney disease and could worsen the progression as well. Despite major reductions in age-adjusted death rates from coronary heart disease and stroke, these continue to be the leading and third most common causes of death, respectively, in the United States. In particular, for every 20 mm Hg increase in systolic blood pressure or 10 mm Hg in diastolic blood pressure, there is a doubling of stroke and coronary artery disease death rates. Kidney Failure related to hypertension continues to grow, especially among the African-American population.

Traditional approaches have mostly included pharmaceuticals targeting different mechanisms that contribute to HTN. However, adequate control of Blood pressure continues to remain a major problem.

Resistant hypertension is defined as blood pressure that remains above goal in spite of the concurrent use of three antihypertensive agents of different classes. Ideally, one of the three agents should be a diuretic and all agents should be prescribed at optimal dose amounts. Patients whose blood pressure is controlled but require four or more medications to do so should be considered resistant to treatment. The prevalence of resistant hypertension is unknown. Cross- sectional studies and hypertension outcome studies suggest, however, that it is not uncommon. In a recent analysis of National Health and Nutrition Examination Survey (NHANES) participants being treated for hypertension, only 53% were controlled to <140/90 mm Hg. In a cross-sectional analysis of Framingham Heart Study participants, only 48% of treated participants were controlled to <140/90 mm Hg and less than 40% of elderly participants (>75 years of age) were at a goal blood pressure.

The benefits of successful treatment, however, are likely substantial as suggested by hypertension outcome studies in general and by the early Veterans Administration cooperative studies, which demonstrated a 96% reduction in cardiovascular events over 18 months with use of triple antihypertensive regimens compared with placebo in patients with severe hypertension (diastolic blood pressure 115 to 129 mm Hg).

Furthermore, as age and obesity are the two most common risk factors for hypertension the prevalence will likely increase as the patient population gets older and heavier. This necessitates development of novel therapeutic approaches to blood pressure control.

Enhanced External Counterpulsation (EECP) is a non-invasive method currently used for the treatment of ischemic coronary disease. During EECP therapy three compressive pneumatic cuffs are wrapped to the calves, lower thighs, and upper thighs. The cuffs inflated sequentially during diastole cause retrograde aortic flow, and increased venous return. During end diastole, the cuffs rapidly deflate, resulting in unloading of the left ventricle and a decrease in systolic blood pressure. In addition there is also evidence that EECP improves endothelial function. Endothelial dysfunction with imbalance of vasodilatory and vasoactive substance is thought to contribute to elevated blood pressure. This leads us believe that EECP, although not used at present for patients with Resistant HTN, may represent a novel, valuable and untapped therapy.

We propose to study the effect of EECP therapy on mean ambulatory blood pressure and noninvasive hemodynamics in subjects with Resistant HTN. We will measure subjects' ambulatory blood pressure and noninvasive hemodynamics parameters at baseline, 4 weeks and 7 weeks. Subjects will undergo a 7 week course (35 sessions) of EECP therapy. Follow up ambulatory BP and non invasive hemodynamic parameters will be measured to evaluate any change in BP.

Our hypothesis is that in patients with Resistant HTN will demonstrate improved Blood pressure after completion of 35 sessions of EECP therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are competent to provide written consent
* Aged 18 to 80 years
* Deemed to be compliant with anti-hypertension medication therapy.
* Subjects with diabetes and/or chronic kidney disease must have a mean systolic blood pressure ≥130 mmHg
* All other subjects must have a mean systolic blood pressure ≥140 mmHg
* Receiving and adhering to full doses of appropriate guideline-recommended antihypertensive drugs from three different classes of antihypertensive agents, including a diuretic
* Female subjects of non-childbearing potential (i.e., post-menopausal for at least 2 years; surgically sterile)
* Deemed to be compliant with anti-hypertension medication therapy

Exclusion Criteria:

* Average sitting systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg
* Known Sleep apnea
* Subjects who have participated in a clinical study involving another investigational drug or device within 4 weeks prior to Screening
* Have hypertension secondary to an identifiable and treatable cause other than sleep apnea
* Acute coronary syndrome < 6 weeks prior to enrollment
* Non-bypassable left main coronary with a luminal stenosis ≥ 50%
* CABG < 3 months or PCI < 6 months prior to enrollment
* Cardiac catheterization < 2 weeks prior to enrollment
* Arrhythmias that would significantly interfere with the triggering of the EECP device.
* Clinically significant valvular heart disease
* Acute myocarditis
* ICD if it has been triggered < 3 months prior to enrollment
* History of deep vein thrombosis, phlebitis, stasis ulcer, pulmonary embolism, and/or aortic aneurysm
* INR ≥ 2.5
* Patients taking over the counter medications that can raise blood pressure, such as

  * Non narcotic analgesics
  * Non steroidal anti-inflammatory agents, including aspirin, Selective COX-2 inhibitors
  * Sympathomimetic agents (decongestants, diet pills, cocaine)
  * Stimulants (methylphenidate, dexmethylphenidate, dextroamphetamine, amphetamine, methamphetamine, modafinil)
  * Alcohol
  * Oral contraceptives
  * Cyclosporine
  * Erythropoietin
  * Natural licorice
  * Herbal compounds (ephedra or ma huang)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean ambulatory 24-hour systolic ambulatory blood pressure | Approximately 50 days

SECONDARY OUTCOMES:
Change from baseline in mean ambulatory 24-hour diastolic ambulatory blood pressure | Approximately 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Darshak H Karia, MD, Principal Investigator — Albert Einstein Medical Center
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States